CLINICAL TRIAL: NCT01691131
Title: Effects of Two Training Protocols in Physical Activity in Daily Life and Balance in Patients With COPD: Land Versus Water
Brief Title: Effects of Two Training Protocols in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Norte do Paraná (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Unopar
Record Dates: First submitted 2012-04-12; First posted 2012-09-24 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: COPD
Keywords: Physical activity in daily life; Balance; COPD; Exercise training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise training on land (Other): High intensity exercise training on land.
  Interventions: Other: Exercise training
- Exercise training on water (Other): High intensity exercise training on water.
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — Comparison of high intensity exercise training on land versus water.
  Other Names: Exercise training on land;; Exercise training on water.

SUMMARY:
Introduction: There is evidence that demonstrate the beneficial effects of pulmonary rehabilitation programs (PR) on symptoms, exercise capacity, muscle strength and quality of life in patients with Chronic obstructive pulmonary disease (COPD). The majority of the studies used high intensity endurance and strength exercise training on land. Exercise on water is an effective form of training that has been used for decades for rehabilitation in different chronic conditions. In addition, there are promising preliminary results on the literature regarding aquatic training in patients with COPD. However, several gaps remain.

Aim: Compare the effects of two rehabilitation programs with 6 months of duration in patients with COPD on physical activity in daily life and balance: land versus water.

Methods: The sample will consist of 36 patients with COPD diagnosed according to the GOLD criteria, 50 years old or more and clinically stable.

Patients will be evaluated in 3 different moments: before the PR, after the PR and 6 months after the end of the PR (follow up). In addition to the assessment of physical activity in daily life and balance, the investigators will also evaluate pulmonary function, peripheral and respiratory muscle strength, body composition, maximal and submaximal exercise capacity, functional status and quality of life.

Both groups (land or water) will be submitted for 3 sessions of exercise training per week, with 45 minutes of duration, during 6 months. The sessions of both groups include the same exercises sequence. Endurance exercise training will be performed on a bicycle and walking on land and strength training using free weights. Workload will be established according to the tests performance on assessment and progression will follow a predetermined schedule and adjusted according symptoms. On water the same approach will be followed.

Expected results: the investigators expect improvement in terms of symptoms, exercise capacity, muscle strength, quality of life, functional status and physical activity in daily life at the end of the two training protocols. However, it is unclear whether one training protocol will be superior than the other. Due to the characteristics involved in the aquatic training, the investigators hypothesized that this type of training can result in better results on balance.

DETAILED DESCRIPTION:
There is evidence that demonstrate the beneficial effects of pulmonary rehabilitation programs (PR) on symptoms, exercise capacity, muscle strength and quality of life in patients with Chronic obstructive pulmonary disease (COPD). The majority of the studies used high intensity endurance and strength exercise training on land. Exercise on water is an effective form of training that has been used for decades for rehabilitation in different chronic conditions. In addition, there are promising preliminary results on the literature regarding aquatic training in patients with COPD. However, several gaps remain.

Therefore, we aim to compare the effects of two rehabilitation programs with 6 months of duration in patients with COPD on physical activity in daily life and balance: land versus water.

The sample will consist of 36 patients with COPD diagnosed according to the GOLD criteria, 50 years old or more and clinically stable.

Patients will be evaluated in 3 different moments: before the PR, after the PR and 6 months after the end of the PR (follow up). In addition to the assessment of physical activity in daily life and balance, the investigators will also evaluate pulmonary function, peripheral and respiratory muscle strength, body composition, maximal and submaximal exercise capacity, functional status and quality of life.

Both groups (land or water) will be submitted for 3 sessions of exercise training per week, with 45 minutes of duration, during 6 months. The sessions of both groups include the same exercises sequence. Endurance exercise training will be performed on a bicycle and walking on land and strength training using free weights. Workload will be established according to the tests performance on assessment and progression will follow a predetermined schedule and adjusted according symptoms. On water the same approach will be followed.

Expected results: the investigators expect improvement in terms of symptoms, exercise capacity, muscle strength, quality of life, functional status and physical activity in daily life at the end of the two training protocols. However, it is unclear whether one training protocol will be superior than the other. Due to the characteristics involved in the aquatic training, the investigators hypothesized that this type of training can result in better results on balance.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis (according to the GOLD criteria);
* Stable condition, no exacerbations or infections in the last 3 months;
* No severe or unstable heart disease;
* No other pathological conditions that could influence the training performance;
* Not have participated in other rehabilitation programs in the last six months.

Exclusion Criteria:

* Occurrence of acute exacerbation during the evaluation period;
* Not understanding or non-cooperation regarding the procedures and research methods;
* Option of the participant to leave the study for any reason;
* Presence of vestibular disorders (BPPV, labyrinthitis, among others).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Physical activity in daily life (measuremet unit: number of steps per day) | four years
  The objectively assessed level of physical activity in daily life will be monitored using the activity monitor Power Walker PW 610 (Yamax, Japan). This device is validated in patients with COPD and the main variables are the number of steps per day and estimation of daily energy expenditure. The monitor will be individually set taking into consideration body weight and step length (measured in a 10-meter walking at usual speed). Patients will wear the device 12 hours per day during 6 days, and the average of these six days will be used for analysis.

SECONDARY OUTCOMES:
Static Balance (Center of Pressure Area in cm2) | four years
  Static balance will be evaluated using a force platform (BIOMEC400, EMG System of Brazil, Brazil), which is a reliable instrument for stabilographic measures in both, older and young adults.
Dynamic Balance (Timed up and go test in seconds) | four years
  Dynamic balance will be assessed by Timed up and go test (TUG).
Exercise capacity (6MWT: distance covered in meters; ISWT: distance covered in meters) | four years
  The 6-minute walking test (6MWT) will be performed to verify functional exercise capacity and the Incremental shuttle walk test (ISWT) to assess maximal exercise capacity.
Quality of life (CRDQ: score in points) | four years
  The Chronic Respiratory Disease Questionnaire (CRDQ) will be applied to assess quality of life.
Functional status (LCADL: score in points) | four years
  Functional status will be assessed by using the questionnaire "London Chest Activity of Daily Living scale" (LCADL). A total score is calculated according to the patient report for each domain.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Pitta, PhD, Study Director — Universidade Estadual de Londrina; Vanessa S. Probst, PhD, Principal Investigator — Universidade Norte do Paraná
Locations (1):
- Universidade Norte do Paraná, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Castro LA, Felcar JM, de Carvalho DR, Vidotto LS, da Silva RA, Pitta F, Probst VS. Effects of land- and water-based exercise programmes on postural balance in individuals with COPD: additional results from a randomised clinical trial. Physiotherapy. 2020 Jun;107:58-65. doi: 10.1016/j.physio.2019.08.001. Epub 2019 Aug 6. PMID 32026836
- [Derived] Felcar JM, Probst VS, de Carvalho DR, Merli MF, Mesquita R, Vidotto LS, Ribeiro LRG, Pitta F. Effects of exercise training in water and on land in patients with COPD: a randomised clinical trial. Physiotherapy. 2018 Dec;104(4):408-416. doi: 10.1016/j.physio.2017.10.009. Epub 2018 Mar 1. PMID 30477678